CLINICAL TRIAL: NCT01605604
Title: Department of Orthopedic Surgery, Faculty of Medicine Siriraj Hospital
Brief Title: Effectiveness of Buddhist Intergrated Group Intervention on Minefulness in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kamolporn Kaewpornsawan, Department of orthopedic surgery, Faculty of Medicine Siriraj hospital, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: si496-2010
Record Dates: First submitted 2012-04-25; First posted 2012-05-25 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: mindfulness EQ adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recieves Buddhist mindfullness (Experimental)
  Interventions: Behavioral: buddhist mind fullness

INTERVENTIONS:
Behavioral: buddhist mind fullness — there are two group one group recieve Buddhist mindfulness group intervention 8 times second group recieve nothing
  Other Names: no other name

SUMMARY:
The pupose of the study is to determine the effectiveness of the Buddhist integrated group intervention improve the mindfulness in adolescents by a randomized controlled trial.The study divede the adolescents in two groups group A recieved the 8 time Buddhist group interventions.Group recieved nothing.The measurement were done pre and post intervention at week1 and week8.The mindfulness score ,the EQ,the MASS score were compared between both groups.

DETAILED DESCRIPTION:
Adolescence behavioural problems are increasing including learning disabilities,game addiction,intolerance etc.The improvement of mindfulness ,the emotional quotient(EQ) proved to be effective to reduce the problems.The original teaching methods in school or in the temple are inadequate from increasing number of adolescent problems. The new technique integrated between Buddhism and group intervention is proposed to improve the mindfulness and EQ in adolescence.

ELIGIBILITY:
Inclusion Criteria:

* adolescents

Exclusion Criteria:

* incomplete qeustionaire and intervention

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The mindfulness score,The EQ score,the MASS score of the participants after intervention. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kamolporn - Kaewpornsawan, M.D., Principal Investigator — Department of orthopaedic surgery Faculty of medicine siriraj hospital Bangkok Thailand
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok, Bangkok, Thailand